CLINICAL TRIAL: NCT04540341
Title: Investigation of the Effectiveness of Mulligan Mobilization Technique and Core Stabilization Exercises in Female Patients With Knee Osteoarthritis: A Randomized Controlled Single-Blind Study.
Brief Title: Effectiveness of Mulligan Mobilization Technique and Core Stabilization Exercise With Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, Meryem BUKE, Research assistant, Pamukkale University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 60116787-020/48052
Record Dates: First submitted 2020-08-27; First posted 2020-09-07 (Actual); Last update posted 2022-04-21 (Actual); Status verified 2022-04

CONDITIONS: Exercise
Keywords: Pain, Joint; Mulligan; Core stabilization
MeSH Terms: conditions — Motor Activity; Arthralgia

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Mulligan mobilization group (Experimental): Painless movement
  Interventions: Other: Mulligan mobilization
- Core stabilization group (Experimental): Abdominal drawing-in maneuver
  Interventions: Other: Core stabilization
- conventional therapy group (Active Comparator): Ultrasound TENS Hotpack
  Interventions: Other: Conventional therapy

INTERVENTIONS:
Other: Mulligan mobilization — Mulligan mobilization technique will be apply.
  Arms: Mulligan mobilization group
Other: Core stabilization — Core stabilization technique will be apply.
  Arms: Core stabilization group
Other: Conventional therapy — Conventional therapy exercise will be apply.
  Arms: conventional therapy group

SUMMARY:
Osteoarthritis (OA) is a chronic disease process characterized by degeneration and inflammation in the joint cartilage and subchondral bone, synovial fluid and joint capsule. One of the most affected joints in OA is the knee joint, and the incidence of OA increases with age.

Different treatment approaches are used in the treatment of osteoarthritis. The aim of the study is to examine the effectiveness of Mulligan technique and core exercises applied to female patients with knee osteoarthritis. In addition, the investigators did not find any study examining the effect of Mulligan technique on static balance in the treatment of OA. This is the secondary aim of the study.

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosed with knee osteoarthritis
* To be in the age range of 40-70
* No lower extremity surgery in the last 6 months.
* Agree to participate in the study

Exclusion Criteria:

* Having had hip-knee replacement surgery
* Surgery planned in the last 6 months
* Having received physical therapy in the last 6 months
* Having uncontrollable hypertension and cardiac problems
* Having been diagnosed with rheumatoid arthritis

Ages: 40 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2020-08-14 (Actual); Primary Completion 2022-02-01 (Actual); Study Completion 2022-04-20 (Actual)

PRIMARY OUTCOMES:
Pain assessment | 10 minutes
  Visual Analog Scale: This scale consists of a straight line with the end points defining extreme limits such as 'no pain at all', which is 0 cm, and 'pain as bad as it could be', which is 10cm.
Range of motion assessment | 10 minutes
  Goniometric measurement
muscle strength assessment | 10 minutes
  by handheld device (Commander Powertrack II brand)
functional level assessment | 5 minutes
  Western Ontario and McMaster Universities Arthritis Index (WOMAC)
aerobic endurance assessment | 6 minutes
  6 minute walk test
balance assessment | 5 minutes
  Stand on one leg test
Timed Up& Go Test | 5 minutes
  Timed Up& Go Test
assessment of quality of life survey | 5 minutes
  Nottingham Health Profile

CONTACTS AND LOCATIONS:
Overall Officials: Meryem Buke, Principal Investigator — Pamukkale University
Locations (1):
- Pamukkale University, Denizli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No